CLINICAL TRIAL: NCT02787655
Title: Aerobic Exercise and Cognitive Training in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B8034-W
Record Dates: First submitted 2016-05-25; First posted 2016-06-01 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Sedentary Lifestyle
Keywords: Aging
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic Exercise + Cognitive Training Group (Experimental): Exercise 3 times a week on a stationary ergometer @ 50-80% of maximal heart rate reserve for 20 minutes to 45 minutes per session; plus 20 minutes of cognitive training using Mindfit program
  Interventions: Behavioral: Aerobic exercise + Cognitive Training Group
- Cognitive Training Only Group (Active Comparator): Cognitive Training Only Group. For this arm of the intervention, randomized participants followed the same guidelines as the cognitive component of the AE+CT group but did not partake in aerobic exercise. To equalize contact/monitoring of the groups this group met for the same total duration time as the AE+CT group; however, instead of aerobic exercise, progressive whole body stretching and toning exercises
  Interventions: Behavioral: Cognitive training Only

INTERVENTIONS:
Behavioral: Aerobic exercise + Cognitive Training Group — stationary bicycling
  Arms: Aerobic Exercise + Cognitive Training Group
Behavioral: Cognitive training Only — 20 minutes of cognitive training using Mindfit program
  Arms: Cognitive Training Only Group

SUMMARY:
The purpose of this study is to examine the impact of a combined cognitive training and aerobic exercise intervention in sedentary older adults. It is hypothesized that the aerobic exercise will potentiate and increase the generalizability of the cognitive training. Importantly, this study will focus on older adults at-risk for mobility disability. This area is of particular importance considering a large percentage of adults are entering old age and therefore likely to suffer from age-related cognitive decline and mobility disability.

To address the investigators' research question 60 adults (age 18-89) will be randomized to one of two 12 week intervention groups: 1) Cognitive Training alone (CT) or 2) Aerobic Exercise + Cognitive Training (AE+CT). The aerobic exercise arm of the study will follow the same format shown to improve a broad range of executive functions in older adults in previous research. The cognitive training arm will consists of a popular commercially-available brain fitness program that has demonstrated specific cognitive improvements and high adherence.

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to examine the impact of a combined cognitive training and aerobic exercise intervention in sedentary older adults. Recent research demonstrated that older adults who participated in aerobic fitness training significantly increased their brain volume. Equally important, the demonstrated enhancement in brain size is related to improvement on specific cognitive tasks. For example, researchers demonstrated that 124 older adults randomly assigned to receive aerobic training experienced substantial improvement in cognitive performance tasks related to speed of processing and working memory. Similarly, neuroimaging studies showed that aerobically trained individuals increased brain activation during various cognitive tasks.

A growing body of research also demonstrates the beneficial effects of cognitive training in later life to promote a healthy brain. For example, researchers demonstrated cognitive interventions targeting memory, reasoning and speed of processing were effective to improve brain function. Unfortunately, despite these promising findings, the generalizability of cognitive training is limited. For example, researchers showed cognitive training tasks designed to improve reasoning, memory, planning, spatial skills and attention in over 11,000 participants demonstrated no transfer effects to untrained tasks, even when the tasks were closely related. The purpose of this study is to see if combing aerobic exercise and cognitive training can enhance the cognitive improvement of each. Specially, the investigators wish to determine if aerobic exercise done immediately before cognitive training can potentiate the improvement.

The investigators hypothesized that the aerobic exercise will potentiate and increase the generalizability of the cognitive training. Importantly, this study will focus on older adults at-risk for mobility disability. This area is of particular importance considering a large percentage of adults are entering old age and therefore likely to suffer from age-related cognitive decline and mobility disability.

Background: Currently the United States has over 23 million Veterans. Of this number, 39.1 percent are over the age of 65 a number that will greatly increase as a large percent of the US population ages. Unfortunately, many of these individuals will suffer from some form of age-related cognitive decline and/or mobility disability. Significantly, declining mental health and mobility disability are primary components of the expected 25 percent growth in health care cost related to the aging crisis in America. And, despite the fact that the United States federal government spends $100 billion dollars annually to cure and/or treat cognitive impairments, successful strategies to improve these impairments remain elusive. The proposed research will substantially advance the development of treatments for cognitive and mobility impairment because the goals explore an intervention that may potentially have pervasive effects on US Veterans quality of life and well-being from a physical as well as a cognitive standpoint.

Methods and Research Plan: To address the investigators' research question 60 adults (age 18-89) will be randomized to one of two 12 week intervention groups: 1) Cognitive Training alone (CT) or 2) Aerobic Exercise + Cognitive Training (AE+CT). The aerobic exercise arm of the study will follow the same format shown to improve a broad range of cognitive functions in older adults in previous research. The cognitive training arm will consists of a popular commercially-available brain fitness program that has demonstrated specific cognitive improvements and high adherence.

Baseline testing will consist of a battery of cognitive function that target verbal fluency, response inhibition, and working memory. Additionally, participant will undergo a structural and functional MRI. Participants will also be evaluated on their physical function as assessed by a 400 meter walk, balance tests, and questionnaires about their daily l functioning. And lastly, all participants will be assessed on their aerobic capacity and for visual outcomes and serum BDNF. Following the 12-week intervention all participants will be post tested in the same manner as the baseline testing.

ELIGIBILITY:
Inclusion Criteria:

* Right handed
* English speaking
* Aged 18 to 89
* Sedentary as defined by < 120 min/week of aerobic exercise over prior 3 months
* Non-demented (MMSE 24)

Exclusion Criteria:

* Severe diabetes requiring insulin
* Cognitive-executive function deficit (MoCA < 26)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe R. Nocera, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nocera J, Crosson B, Mammino K, McGregor KM. Changes in Cortical Activation Patterns in Language Areas following an Aerobic Exercise Intervention in Older Adults. Neural Plast. 2017;2017:6340302. doi: 10.1155/2017/6340302. Epub 2017 Mar 6. PMID 28367334

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aerobic Exercise + Cognitive Training Group | Cognitive Training Only Group
Started | 40 | 38
Completed | 29 | 26
Not Completed | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Aerobic Exercise + Cognitive Training Group: Randomized participants attended exercise training sessions and cognitive training sessions
- Cognitive Training Only Group: Participants will follow the same guidelines as the cognitive component of the AE+CT group but did not partake in aerobic exercise.
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise + Cognitive Training Group | Cognitive Training Only Group | Total
Number analyzed (Participants) | 40 | 38 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 40 | 38 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (6.34) | 72.09 (6.43) | 71.24 (6.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 10 | 25
  White | 25 | 28 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 38 | 78

OUTCOME MEASURES:

1. Primary Outcome: Change Executive Language Functions (Category Verbal Fluency)
Description: The Category Verbal Fluency Test is demonstrated to be reliable and valid among adults aged 50 to 89. For Category Verbal Fluency, participants are asked to generate words from a category (e.g., colors) within 60 seconds. A higher change score represents better performance on the outcome.
Time Frame: change from pre and post separated by 12 weeks
Measure: Mean (Standard Deviation); unit: Number of Fluent Words within 60 seconds
Arm/Group | Aerobic Exercise + Cognitive Training Group | Cognitive Training Only Group
Number analyzed (Participants) | 29 | 26
Number of Fluent Words within 60 seconds | 5 (2.5) | -1 (4)

ADVERSE EVENTS:
Time Frame: From baseline through the 12 week intervention concluding once all post testing was completed.
Arm/Group | Aerobic Exercise + Cognitive Training Group | Cognitive Training Only Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 0/40 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT02787655/Prot_SAP_000.pdf